CLINICAL TRIAL: NCT07188363
Title: Prospective Follow-up Study of Patients Undergoing Ankle Ligament Surgery
Brief Title: French Ankle Ligament Surgery Cohort Study
Acronym: AnkleCDS
Status: Recruiting | Type: Observational
Sponsor: Chirurgie Du Sport (Other)
Responsible Party: Principal Investigator, HARDY Alexandre, Surgeon, Chirurgie Du Sport
Other Study IDs: AnkleCDS
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Ankle (Ligaments); Instability (Old Injury); Ankle Ligament Rupture; Ankle Instability; Syndesmotic Injury
Keywords: ankle; ligamentoplasty; surgery; orthopedy; FHL; rupture; ligament; syndesmosis; instability; retensioning; flexor hallucic longus
MeSH Terms: conditions — Ankle Injuries; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ligament reconstruction — Retensioning involves restoring the tension in a ligament or soft tissue that has become lax, often due to injury or joint instability. This technique is typically used for ligaments that do not require complete reconstruction but have lost their functional tension. Ligament reconstruction is a surgical procedure to replace or repair a damaged ligament, often using grafts (autografts or allografts). It aims to restore joint stability and function, particularly in cases of significant ligament damage or rupture. Syndesmosis surgery involves repairing or reconstructing the fibrous joint between two bones (e.g., the tibia and fibula). It may involve screw fixation, suture-button devices, or grafts to restore the alignment and stability of the syndesmosis.
  Other Names: Syndesmosis; Retensioning

SUMMARY:
This 20-year cohort study foolows patients after ankle ligament reconstruction surgery to evaluate re-rupture rates, long term functional outcomes, return to sport rates ans complications? The goal is to provide insights into the procedure's durability and effectiveness to enhance patient care.

DETAILED DESCRIPTION:
This study is a long term cohort analysis involving patient who have undergone ankle ligament reconstruction surgery (ligamentoplasty). The goal is to follow these patients over 20 year period to assess several important outcomes. Specifically, the study aims to evaluate the rate of re-ruptures, the rates and quality of return to sport, long term functional outcomes using validated scoring systems and the incidence of complications related to the procedure.

By collecting detailed and consistent data over two decades, the research seeks to provide valuable insights into the durability and effectiveness of ankle ligament reconstruction surgery, contributing to a better understanding and improved care for patients

ELIGIBILITY:
Inclusion Criteria:

* Retensioning, ankle ligament reconstruction or syndesmosis repair surgery

Exclusion Criteria:

* Patient refusal

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled ine the Ankle CDS cohort by one of the surgeons of the Chirurgie du Sport and meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2042-08-30 (Estimated); Study Completion 2062-08-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of a ligament tear | From the surgery to the end of the study (20years of follow-up for each patient)

SECONDARY OUTCOMES:
Return to sport | From the surgey to the end of follow up (20 years)
  Return to sport after surgery with the level of return, the type of sport and the delay.
  Questions regarding the return to sport at 6 months, 1 year, 2 years and every 2 years
Visual Analogue Scale | From the surgery to the and of the follow-up (20 years for each patient)
  The VAS score (Visual Analogue Scale) is a simple and widely used method for assessing subjective experiences, such as pain intensity, fatigue, or discomfort. It typically consists of a horizontal or vertical line, usually 10 cm in length, with endpoints representing the extremes of the experience being measured: 0: "No pain" (or "no discomfort"). 10: "Worst pain imaginable" (or "maximum discomfort") Evaluated during the 3 first days after surgery, at 6 months, 1 year, 2 years and every 2 years
Ankle Ligament Reconstruction - Return to Sport Injury score | From the surgery to the end of foolow-up (20 years for each patient)
  The ALR-RSI (Ankle Ligament Reconstruction - Return to Sport Injury) score is used to assess the patient's psychological state and apprehension regarding their return to sports activities. The score ranges from 0% (the lowest level of psychological readiness) to 100% (the highest level of psychological readiness). Questionnairy at 6 months, 1 year, 2 years and every 2 years
Foot and Ankle outcome score | From the surgey to the end of follow-up (20 years of follow-up for each patient)
  Foot and Ankle outcome score is used to evaluate the patient's functional abilities, symptoms, and quality of life related to ankle and foot conditions. The FAOS (Foot and Ankle Outcome Score) is a 42-item questionnaire comprising five subscales: pain (9 items), other symptoms (7 items), activities of daily living (ADL) (17 items), sports/recreation (5 items), and quality of life (4 items). Each question is rated on a 5-point Likert scale (none, mild, moderate, severe, and extreme problems) from 0 to 4. The score for each subscale is calculated by summing all the individual scores within the subscale and dividing the result by the maximum possible score for that subscale. The normalized score is then converted to a scale of 0 to 100, where 100 indicates no problems and 0 indicates severe problems. Measured at 6 months, 1 year, 2 years and every 2 years.
Cumberland Ankle Instability Tool (CAIT) | From the surgery to the end of the follow-up (20 years for each patient)
  The questionnaire consists of 9 questions that the patient answers independently, evaluating ankle pain, subjective instability during activities such as running or hopping, and the ankle's ability to handle twisting episodes. The responses to the nine questions are summed to produce a total score ranging from 0 to 30 points. A higher score indicates better ankle stability. Measured at 6 months after surgery, 1 year, 2 years and every 2 years
Foot an Ankle Ability Measure | From the surgery to the end of follow-up (20 years for each patient)
  Foot and Ankle Ability Measure (FAAM) is a tool designed to assess a patient's functional abilities and symptoms specifically related to their foot and ankle during daily activities and sports. It consists of two subscales: Activities of Daily Living (ADL): 21 items. Sports: 8 items. Each item is rated on a 5-point Likert scale: 4 = No difficulty 3 = Slight difficulty 2 = Moderate difficulty 1 = Extreme difficulty 0 = Unable to perform Scoring : Add the scores for all items within the subscale to calculate the total item score. Multiply the total number of answered items by 4 to determine the highest potential score (e.g., 84 for ADL and 32 for Sports if all items are answered). Divide the total item score by the highest potential score and multiply by 100. This gives the FAAM score, which ranges from 0% (lowest function) to 100% (highest function). Interpretation : A higher score indicates a greater level of physical function.
  Measured at 6 months, 1 year, 2 years and every 2 years
Complications | From the surgery to the end of follow-up (20 years for each patient)
  Complications of the surgery recorded or re-operations : - Removal of hardware - Infection -Hematoma -Further ankle stabilization -Cartilage surgery -Arthrodesis -Ankle prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Hardy, MD, Principal Investigator — Chirurgie Du Sport
Locations (1):
- Chirurgie du Sport, Paris, Paris, France